CLINICAL TRIAL: NCT06790901
Title: EVALUATION of PEROPERATIVE ATELECTASIS with LUNG ULTRASOUND SCORE in GENERAL ANAESTHESIA MAINTENANCE METHODS
Brief Title: Effects of Anesthesia on Atelectasis
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Oguzhan Karayaka, MD, Zonguldak Bulent Ecevit University
Other Study IDs: 2023/16-6
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Atelectasis; General Aneshesia
Keywords: Lung Ultrasound Score; general anesthesia; Atelectasis; Inhalation agents
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group Total IV anesthesia
  Interventions: Procedure: LUNG ULTRASOUND
- Group Sevoflurane
  Interventions: Procedure: LUNG ULTRASOUND
- Group Desflurane
  Interventions: Procedure: LUNG ULTRASOUND

INTERVENTIONS:
Procedure: LUNG ULTRASOUND — Determination of atelectsis By Lung Ultrasound Score

SUMMARY:
We know that respiratory functions of patients are affected under general anaesthesia. Although there are many underlying causes of ventilation-perfusion mismatch in the airways, the main cause is atelectasis during general anaesthesia.

Atelectasis occurs in almost all patients receiving general anaesthesia. The main cause of atelectasis is the loss of muscle tone during general anaesthesia. Postoperative atelectasis was described in the last century. It is defined as the closure of the alveoli due to a decrease in inspiratory force and collapse of the lung and the resulting loss of aeration.

Inhalation anaesthetics have been shown to cause hypoxic pulmonary vasoconstriction in studies. However, not all inhalation anaesthetics affect the airways in the same way.

In patients who will undergo surgical procedures under different general anaesthesia maintenance methods, conditions that disrupt the ventilation-perfusion balance in the lung peroperatively can be diagnosed and monitored early, easily and inexpensively by lung ultrasonography.

Lung ultrasound is a noninvasive, reliable, reliable, radiation-free imaging method that provides instantaneous imaging at the bedside. Lung ultrasound score is a scoring system that provides scoring of the loss of ventilation in the lung. For this purpose, it was aimed to divide both lung tissues into 12 areas and to give a score between 0 and 3 points and to show the severity of the loss of aeration according to the resulting total score.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old ASA I-II Surgical procedure time between 2 hours and 5 hours in supine position Patients who will undergo rhinoplasty, septorhinoplasty operation Patients whose consent was obtained with an informed consent form

Exclusion Criteria:

* Those with a history of malignant hyperthermia,
* People with alcohol or drug addiction,
* Presence of dementia or confusion,
* Uncooperative patients,
* Those with respiratory disease,
* Those with coronary artery disease, congestive heart failure,
* Patients with unstable blood pressure,
* Significant anaemia, liver or kidney disease,
* Women during pregnancy or lactation,
* Allergy to anaesthetic agents,
* Body mass index (BMI) >30 kg/m2,
* Those with sepsis or bacterial infection, Body temperature below 35°C and above 38°C at control value

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-65 years old, ASA I-II, who will undergo rhinoplasty, septorhinoplasty operation
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Peroperative Atelectasis | from induction to postoperative 1st hour

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguladk Bulent ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No